CLINICAL TRIAL: NCT02124369
Title: Pancreatic Resectability in Cancers With Known Limited Extension (PRICKLE) - A Single-centre Phase 2a Study of Gemcitabine Plus Nab-paclitaxel for Borderline Unresectable Locally Advanced Pancreatic Cancer
Brief Title: Pancreatic Resectability in Cancers With Known Limited Extension (PRICKLE)
Acronym: PRICKLE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Cancer Research UK (Other); Celgene (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Dr Bristi Basu, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRICKLE; 2013-004200-19 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-28 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic cancer; locally advanced; unresectable
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abraxane & gemictabine (Other): Abraxane, IV, 125mg/m2 and gemcitabine, IV, 1000mg/m2, on days 1,8 & 15 per 28 day cycle, up to a maximum of 6 cycles.
  Interventions: Drug: Abraxane; Drug: Gemcitabine

INTERVENTIONS:
Drug: Abraxane — 125mg/m2, IV, on days 1,8 & 15 of each 28 day cycle, up to 6 cycles.
  Other Names: nab-paclitaxel
Drug: Gemcitabine — 1000mg/m2, IV, on days 1,8 & 15 of a 28 day cycle, up to 6 cycles.
  Other Names: Gemzar

SUMMARY:
Pancreatic cancer is difficult to treat, and even in a situation where an operation can be performed to remove the cancer, the disease can unfortunately come back soon afterwards. When pancreatic cancer is more advanced, the outcomes are even less positive. Recently, a large international study showed that combining a chemotherapy drug that is standard for treating pancreatic cancer, called gemcitabine with a new chemotherapy drug called Abraxane was more effective than gemcitabine alone for patients with advanced pancreatic cancer.

The purpose of this study is to determine whether this combination of gemcitabine and Abraxane can shrink a pancreatic cancer that is not thought to be operable enough to enable it to be removed by surgery. It is hoped that in this way, the treatment may improve the outcome. In addition, in this study we would like to analyse the appearances of the tumour using imaging, and collect blood and tumour samples to try to confirm laboratory research that has been carried out with this treatment.

DETAILED DESCRIPTION:
This is a single-centre, non-randomised, phase 2a, single arm, Simon two-stage design trial of nab-paclitaxel and gemcitabine (ABX/GEM) in patients with histological documentation of pancreatic ductal adenocarcinoma (PDAC) who are determined by central radiological review to have "category 2" borderline unresectable LAPC. We will investigate the feasibility of administering ABX/GEM in terms of safety and efficacy, and will study activity both in terms of radiological response and the feasibility of downstaging patients to "category 1" status, in order to attempt resection after up to 6 cycles of combination treatment. In addition to adding to data on the safety and tolerability of this combination, peri- and post-operative morbidity following this treatment will be evaluated. As part of the trial, detailed correlative studies will be undertaken to evaluate the mechanism of action of the combination, at a tissue level, a circulating biomarker level and a radiological level.

We propose that the tumour shrinkage (response) seen in Stage IV pancreatic cancer patients as a result of ABX/GEM may translate to a realistic prospect of downstaging borderline unresectable LAPC tumours sufficiently to enable resection. Notionally, even in the absence of a classical partial response by RECIST criteria (≥30% reduction in sum of longest diameters) a beneficial outcome may arise from any tumour shrinkage sufficient to permit the tumour to be separated from major vessels thus rendering it resectable. Such an outcome may significantly alter the poor survival outcomes in this group of patients. The PRICKLE clinical study paradigm is useful for evaluating novel agents and combinations that show impressive activity in the pre-clinical or advanced setting and offers an opportunity for detailed correlative translational studies to evaluate activities of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with borderline unresectable advanced pancreatic adenocarcinoma, defined as Category 2 by central radiological review.
* Aged 18 years or over at the time of signing the informed consent form.
* Documented histological or cytological diagnosis of pancreatic ductal adenocarcinoma.
* ECOG performance status 0-1.
* Life expectancy of at least 12 weeks.
* Willing and able to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Adequate haematological function defined by:
* Absolute neutrophil count (ANC) ≥1,500 cells/mm3 (1.5 x 109/L).
* Haemoglobin ≥8.0 g/dL (80 g/L) (may be increased to this level with transfusion as long as there is no evidence of active bleeding).
* Platelets ≥100x 109/L
* Adequate renal function defined by serum creatinine≤1.5 x ULN or calculated creatinine clearance by Cockcroft-Gault of ≥50 ml/min.
* Adequate hepatic function defined by:
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN)
* Total bilirubin ≤1.5 x ULN
* Patients may have endoscopic or radiologic stenting to treat biliary obstruction. If so, bilirubin must return to ≤1.5 x ULN prior to enrolment.
* Received no prior therapy for their disease.
* Measurable disease by RECIST 1.1 criteria. Tumour assessments and measurements must be done within 28 days before the patient receives the first dose of ABX/GEM.
* All Women of Child Bearing Potential (WoCBP) and all sexually active male patients must agree to use effective contraception methods throughout the study and for 6 months after the final dose of trial drug.

Exclusion Criteria:

* Patients with metastatic PDAC, or disease which is amenable to resection with curative intent. These include tumours which are defined as Category 1 or 3 by central radiological review.
* Other invasive malignancies diagnosed within the last 5 years, with the exceptions of adequately treated localized cured prostate cancer, in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for three years or more and are deemed at negligible risk for recurrence, are eligible for the trial.
* Known allergy or hypersensitivity to ABX or GEM.
* Routine use of oral anti-oxidant supplements: beta-carotene, selenium, lutein, zeaxanthin, lycopene, pycnogenol, fernblock, omega-3S, vitamin C, vitamin E, astaxanthin. If recent use, a washout period of 5 half-lives is required.
* Patients with pre-existent ischemic heart disease particularly those under active treatment for coronary disease, will be excluded from Sonuvue dynamic contrast enhanced ultrasound investigation due to sporadic reports of cardiac ischemia in this population. They will be eligible for the rest of the study, as long as their cardiac status does not preclude surgery.
* Significant acute or chronic medical or psychiatric condition, disease or laboratory abnormality which in the judgment of the Investigator would place the patient at undue risk or interfere with the study. Examples include, but are not limited to:
* Patients who have had a venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation who are not appropriately anti-coagulated or have had a NCI CTCAE (version 4.0) Grade 2 or greater bleeding episode in the 4 weeks before Day 1.
* Patients taking warfarin, unless it is possible for the patient to be switched to a low molecular weight heparin for the duration of the study
* Patients with a significant history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months.
* Cirrhotic liver disease, ongoing alcohol abuse, or known chronic active or acute hepatitis B, or hepatitis C.
* Known infection with HIV.
* Women, who are pregnant, plan to become pregnant or are lactating (during the study or for up to 6 months after the last dose).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Tumour resection rate | 18 months
  Is the combination of ABX/GEM effective in shrinking LAPC tumours sufficiently to permit resection.

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 18 months
  Determining the causality of Adverse Events and Serious Adverse Events

OTHER OUTCOMES:
Radiological response by percentage change | 18 months
  Radiological response as determined by percentage change in sum of longest diameters for all target lesions at 3 or 6 months from the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristi Basu, Dr, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom

REFERENCES:
- See also: Pancreatic Cancer UK — http://www.pancreaticcancer.org.uk/
- See also: CancerHelp UK from Cancer Research UK — http://www.cancerresearchuk.org/cancer-help/
- See also: Cancer Backup — http://www.macmillan.org.uk/home.aspx
- See also: Macmillan Cancer Support — http://www.macmillan.org